CLINICAL TRIAL: NCT01339325
Title: Laparo-endoscopic Single Site Cholecystectomy Versus Standard Laparoscopic Cholecystectomy
Brief Title: Laparo-endoscopic Single Site (LESS) Cholecystectomy Versus Standard LAP-CHOLE
Acronym: LESSCHO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: San Giovanni Addolorata Hospital (Other)
Responsible Party: Marco Maria Lirici, San Giovanni Addolorata Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGAddolorataH-MLirici-14-93
Record Dates: First submitted 2011-03-30; First posted 2011-04-20 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-03

CONDITIONS: Cholelithiasis
Keywords: Laparo-endoscopic single site cholecystectomy; Quality of Life; Postoperative Pain; Cosmetics; Complication
MeSH Terms: conditions — Cholelithiasis; Pain, Postoperative | interventions — Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LESS cholecystectomy (Active Comparator): Laparo-endoscopic single site cholecystectomy, the entire surface of the patient's abdomen is covered by plaster at the end of the operation. Patient does not know which kind of procedure he underwent before discharge.
  Interventions: Procedure: Cholecystectomy
- Standard LAP-CHOLE (Active Comparator): Standard laparoscopic cholecystectomy. The entire surface of the patient's abdomen is covered by plaster at the end of the operation. Patient does not know which kind of procedure he underwent before discharge.
  Interventions: Procedure: Cholecystectomy
- LESS Cholecystectomy not blind (Active Comparator): Laparo-endoscopic single site cholecystectomy. The patient is aware of the procedure he underwent.
  Interventions: Procedure: Cholecystectomy

INTERVENTIONS:
Procedure: Cholecystectomy — Standard laparoscopic cholecystectomy The first cannula is inserted with an "open laparoscopy" technique. LCs are performed with either HF or US energized dissection, standard or fundus-first gallbladder dissection, closure of the artery by ligature/clip or US, closure of cystic duct by ligature/clip.
  Laparo-endoscopic single site cholecystectomy
  The TriPort device is inserted at the navel site through a 15 to 25 mm incision with an "open laparoscopy" technique. Two working instruments are inserted (one grasper and one energised device) through the TriPort. A further 1.8 or 3 mm instrument inserted through the larger gel valve, parallel to a 5 mm dissecting instrument, is used in some cases to enhance exposure. Gallbladder dissection is accomplished either after preparation of the cystic duct and artery or with a fundus-first technique, by means of HF electrosurgery or US shears.The cystic artery is divided between clips or by US scissors. The duct is divided between clips.

SUMMARY:
The aim of this study is to assess possible differences between the LESS approach and the standard laparoscopic approach to cholecystectomy. In particular, the Postoperative Quality of Life (QoL) will be investigated by analyzing the followings: length of hospital stay (LoS), postoperative pain, cosmetics and the results of SF 36 questionnaire. Furthermore, operative time, conversion to standard LC rate, difficulty of exposure, difficulty of dissection, and complication rate will be compared.

DETAILED DESCRIPTION:
The aim of this study is to assess possible differences between the LESS approach and the standard laparoscopic approach to cholecystectomy. In particular, the Postoperative Quality of Life (QoL) will be investigated by analyzing the followings: length of hospital stay (LoS), postoperative pain, cosmetics and the results of SF 36 questionnaire. Furthermore, operative time, conversion to standard LC rate, difficulty of exposure, difficulty of dissection, and complication rate will be compared.

Altman nomograms were used to calculate the presumed sample size of an actual RCT, arbitrarily assuming a most likely small standardized difference (0.3). With a significant criterion set at 0.05, using a two-tailed test, the number of patients per group, required to have a 90% power is ~500. Therefore, it was decided to carry on a pilot trial, enrolling 40 patients (20 each group), to assess differences in any of the end-points and tailoring the sample size of the larger multicenter RCT accordingly.

This dual-institutional prospective, randomized pilot trial was conducted during 2009 obtaining information on the power and sample size needed for a planned multicenter randomized control trial. Our results showed that Quality of life data concerning LESS cholecystectomy are somewhat controversial: cosmetics and SF36 role emotional parameter significantly improved, no differences were found in length of hospital stay, early postoperative pain (same day of surgery) was higher but no impact on need for pain-relieving medications was found. Altman nomograms were used again to calculate the presumed sample size of an actual RCT based on the differences found on our initial results. With a significant criterion set at 0.05, using a two-tailed test, the number of patients per group, required to have a 90% power in this multicenter RCT is ~180 patients.

Study design Randomization is performed preoperatively and stratification is performed intraoperatively, after visualization of the operative field. Patients are randomized to one of three groups: LESS cholecystectomy blind, standard LC, LESS cholecystectomy not blind. Patients are stratified into 3 groups: Nassar grade I, II, III, according to the grade of difficulty of cholecystectomy (Nassar score) assessed at the initial inspection of the operating field.

Patients of the first two groups do not know the treatment received until their discharge. A large drape is used to cover the abdomen after surgery, thus hiding the surgical wounds. Patients of the LESS cholecystectomy not blind group are aware of the procedure they undergo. The third arm is intended to better evaluate the influence of psychological factors on postoperative pain, cosmetics and quality of life.

All operations are performed by high-skilled laparoscopic surgeons (one each institution) with over 15-year experience in advanced laparoscopic surgery.

Difficulty (impaired) of exposure and difficulty of dissection are assessed subjectively by the operating surgeon and scored 1 to 4, being 1 "no difficulties", 4 "the most difficult" with need for conversion.

Perioperative care is similar in all patients and in all institutions. An independent physician will assess the patient postoperatively in each institution. Postoperative pain is evaluated with a visual analogue scale (VAS) from 1 to 10, with 1 being "the least" pain, 10 "the most" pain, on the day of surgery, on postoperative day 1, 2 (discharge) and at 1-month follow-up. Pain is also deduced from the assumption of pain relieving medications. Patients will receive pain medications only on demand and these will be given in incremental strength beginning with peripheral analgesics as Non-Steroidal Anti-Rheumatic agents (NSAR).

Individual satisfaction for the cosmetic result is evaluated with a visual analogue scale (VAS) from 0 to 100% with 0 being "the worse" result, 100 "the best" one. Cosmetics is also evaluated by measuring the length of umbilical incision at the end of the operation in all study groups. The incision length is measured after gallbladder removal (during standard LC the incision may be enlarged to allow the passage of thick gallbladder or bigger stones).

QoL is assessed at the time of surgery and further assessed at postoperative month 1 by the SF36 questionnaire.

Randomization Randomization is performed preparing three sets of 30 numbered, opaque, sealed envelopes, the envelops of each set containing indications for 10 LESS cholecystectomies, 10 standard LC and 10 LESS cholecystectomies not blind. One set of envelopes is kept at each involved Institution. The envelopes are opened in numeric order for each patient by an assistant not involved in the surgical operations, right before surgery. The surgeons perform a standard LC or a LESS cholecystectomy (blind or not blind) as indicated on the sheet inside the envelopes.

Data analyses Data are analysed using the software XLSTAT Version 2009.5.01 (Addinsoft). An "intent-to-treat" analysis will be performed.

Patients demographics across the treatment groups are compared by chi-square test for categorical measures, and by t-test for continuous data. Mann-Whitney U test is used to compare LoS, postoperative pain VAS, cosmetics VAS, length of skin incision, 8 parameters of SF36, operating time, difficulty of exposure, difficulty of dissection in the two arms. Chi-square test is used to compare conversion rate and administration of pain medication, which is dichotomized as yes or no, in the three arms. All variables are significant at p< 0.05. Logistic model results are reported as odds ratios, two-sided 95% confidence intervals, and p values.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75
* BMI < 35
* no previous upper GI or right colonic surgery with severe adhesions gallstones with absence of clinical signs of acute cholecystitis, bile duct stones or pancreatitis.
* ASA I-III
* Nassar grade of difficulty in performing a laparoscopic cholecystectomy I-III
* diagnosis: cholelithiasis

Exclusion Criteria:

* cholecystitis
* existence of common duct stones
* presence of biliary cancer
* Previous abdominal surgery on organs of the supramesocolic space

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative Quality of Life (QoL) | one month
  Postoperative Quality of Life (QoL) will be the primary endpoint: QoL will be assessed analysing the followings: length of hospital stay (LoS), postoperative pain, cosmetics and the results of SF 36 questionnaire.

SECONDARY OUTCOMES:
operative time | day 1
  operative time is expressed in minutes from the first skin incision on the patient's abdomen to the closure of the last laparoscopic incision
conversion rate to standard LC | day 1
  Conversion rate is intended:
  for the two single access laparoscopic cholecystectomy arms as the number and percentage of procedures during which one or more laparoscopic cannulas are introduced to accomplish surgery or a laparotomy is required.
  for the standard laparoscopic cholecystectomy arm as the number and percentage of procedure during which a laparotomy is required to accomplish surgery.
surgeon perception of difficulty of exposure measured with a Visual Analog Scale (VAS) with 0 to the least difficult and 5 to the most difficult | day 1
surgeon perception of difficulty of dissection measured with a Visual Analog Scale (VAS) with 0 to the least difficult and 5 to the most difficult | day 1
complication rate | one month
  complications are divided into intraoperative and postoperative complications. Intraoperative complications rate is the rate of the following complications that may occur intraoperatively in all 3 study groups: bleeding, bile duct injuries, visceral injuries, gallbladder rupture.
  Postoperative complications rate is the rate of the following complications that may occur within 1 month in all 3 study groups: bleeding, intra-abdominal fluid collection, pancreatitis, bile duct injury, pain caused by missed CBD stones, infection of the skin incision/s, incisional hernia.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Maria Lirici, FACS, Principal Investigator — San Giovanni Hospital
Locations (1):
- San Giovanni Hospital, Rome, Lazio, Italy

REFERENCES:
- [Derived] Steinemann DC, Raptis DA, Lurje G, Oberkofler CE, Wyss R, Zehnder A, Lesurtel M, Vonlanthen R, Clavien PA, Breitenstein S. Cosmesis and body image after single-port laparoscopic or conventional laparoscopic cholecystectomy: a multicenter double blinded randomised controlled trial (SPOCC-trial). BMC Surg. 2011 Sep 12;11:24. doi: 10.1186/1471-2482-11-24. PMID 21910897